CLINICAL TRIAL: NCT07388381
Title: Superficial Vein Thrombosis of the Upper Limb in Bacteremia Associated With PICCline and Midline Catheters: Frequency and Clinical Consequences
Acronym: THROMBI-CATH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 25-PP-07
Record Dates: First submitted 2026-01-23; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Catheter Associated Infection
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Catheter Associated Infection (Experimental)
  Interventions: Other: Follow-up for catheter-related bacteremia

INTERVENTIONS:
Other: Follow-up for catheter-related bacteremia — Clinical follow-up and outcomes of patients with catheter-related bacteremia

SUMMARY:
The use of long-term peripheral venous catheters inserted in the upper limb (PICC lines and Midlines) has increased markedly over recent years.

Catheter-related bacteremias and venous thromboses are the main complications associated with these catheters. These events may occur independently or simultaneously. In addition, venous thromboses may involve the superficial venous system (SVT) or the deep venous system (DVT).

Current guidelines define septic thrombophlebitis as the association of a bacteremia and a DVT along the venous course of the catheter. This represents a severe complication of catheter-related bacteremia, leading to a modification in the duration of antibiotic therapy. However, SVTs associated with catheter-related bacteremias along the catheter pathway are not included in the definition of septic thrombophlebitis and are not addressed by specific recommendations.

The objective of this study is therefore to assess the impact of upper-limb SVT on the frequency of unfavorable outcomes in catheter-related bacteremias related to PICC and Midline catheters, in order to determine whether superficial venous thrombosis occurring in the context of a catheter-related bacteremia should be considered a distinct entity not falling under the diagnosis of septic thrombophlebitis (and therefore not requiring a modification of antibiotic treatment duration, in accordance with current guidelines), or whether, conversely, it should be considered equivalent to septic thrombophlebitis, as is the case for deep venous thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalization in a department of Nice University Hospital
* Expected length of hospitalization ≥ 72 hours
* Diagnosis of catheter-related bacteremia on PICCline or Midline.
* Affiliation with a social security system
* No objection to the study

Exclusion Criteria:

* Pregnant or breastfeeding women
* Legal protection measures (patients under guardianship, trusteeship, or judicial protection)
* Inability to remove the catheter
* Doppler ultrasound showing DVT in the upper limb at selection.
* Inability to perform the initial routine Doppler ultrasound
* Withdrawal of the patient's consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of unfavorable outcomes according to the presence or absence of superficial venous thrombosis (SVT) | At day 28 after completion of treatment for catheter-related bacteremia
  An unfavorable outcome is defined as a composite endpoint including at least one of the following:
  * Relapse of bacteremia documented with the same microorganism and/or
  * Extension of superficial venous thrombosis to the deep venous system (deep vein thrombosis and/or pulmonary embolism) and/or
  * Infectious complications related to the initial diagnosis of catheter-related bacteremia, including infective endocarditis, deep abscess, septic thrombophlebitis, osteoarticular infection, or any other complication related to CRBSI, and/or
  * Septic shock.

SECONDARY OUTCOMES:
Describe the risk factors associated with the occurrence of deep vein thrombosis. | At day 28 after completion of treatment for catheter-related bacteremia
  Comparison of patient parameters and management with the course of catheter-related bacteremia
Describe the imaging findings and the evolution of catheter-related deep vein thrombosis | At day 14 after completion of treatment for catheter-related bacteremia
  Comparison of echo-doppler imaging between inclusion and 14 days after antibiotics treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, CHU de Nice, France

IPD SHARING:
Plan to Share IPD: No